CLINICAL TRIAL: NCT01992809
Title: Polyunsaturated Fatty Acid (Pufa) Omega 3 in the Reduction of the Inflammatory Component of the Nonalcoholic Steatohepatitis (Nash):Randomized Placebo Controlled Study
Brief Title: Omega 3 Supplementation in Fatty Liver
Acronym: OMEGA 3 NASH
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Claudia Pinto Marques Oliveira, PhD, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 0681/09CAPPESQ
Record Dates: First submitted 2013-11-07; First posted 2013-11-25 (Estimated); Last update posted 2013-11-25 (Estimated); Status verified 2013-11

CONDITIONS: Fatty Liver
Keywords: Nonalcoholic fatty liver; omega 3
MeSH Terms: conditions — Fatty Liver; Non-alcoholic Fatty Liver Disease | interventions — Docosahexaenoic Acids

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Omega 3 (Active Comparator): Omega-3 group (n=30) received capsules containing 945 mg of Omega-3 PUFA [α linolenic acid/ 64%, eicosapentaenoic acid (EPA)/16% and docosahexaenoic acid (DHA)/21%], in 3 capsules/ day
  Interventions: Dietary Supplement: Omega 3
- placebo mineral oil (Placebo Comparator): placebo mineral oil 3 ml/day

INTERVENTIONS:
Dietary Supplement: Omega 3 — Omega-3 group (n=30) received capsules containing 945 mg of Omega-3 PUFA [α linolenic acid/ 64%, eicosapentaenoic acid (EPA)/16% and docosahexaenoic acid (DHA)/21%], in 3 capsules/ day
  Arms: Omega 3

SUMMARY:
Nonalcoholic fatty liver disease (NAFLD) is a clinical and pathological condition, whose spectrum can range from steatosis to steatohepatitis and cirrhosis, in patients without a history of alcohol abuse. Nonalcoholic steatohepatitis (NASH), the severe form of (NAFLD), has emerged as a clinically important type of chronic liver disease in industrialized countries and is characterized pathologically by hepatocellular ballooning, Mallory's hyaline, scattered inflammation and perisinusoidal fibrosis. NASH associated with cirrhosis can decompensate into subacute liver failure, progress to hepatocellular cancer and reoccur post transplantation.In the absence of established treatment, therapy is generally directed to treatment of risk factors for metabolic syndrome. Recently, some studies have been demonstrated that Polyunsaturated fatty acids (PUFAs), omega3 type, could reduced TNFalfa, IL6, aminotransferases, insulin resistance and steatosis verified by ultrasound. Neverthless, this is the first study that evaluate liver histology after six months of PUFA (omega3) in the treatment of patients with NASH.

DETAILED DESCRIPTION:
Nonalcoholic fatty liver disease (NAFLD) is a clinical and pathological condition, whose spectrum can range from steatosis to steatohepatitis and cirrhosis, in patients without a history of alcohol abuse. Nonalcoholic steatohepatitis (NASH), the severe form of (NAFLD), has emerged as a clinically important type of chronic liver disease in industrialized countries and is characterized pathologically by hepatocellular ballooning, Mallory's hyaline, scattered inflammation and perisinusoidal fibrosis. NASH associated with cirrhosis can decompensate into subacute liver failure, progress to hepatocellular cancer and reoccur post transplantation.

The 'two-hit' hypothesis has been proposed to explain the pathogenesis of NASH, with an initial metabolic disturbance (insulin resistance) causing steatosis and a second pathogenic stimulus promoting oxidative stress, increased generation of reactive oxygen species (ROS), lipid peroxidation, and resultant NASH . Insulin resistance plays a major role in hepatic fat accumulation through increased influx of free fatty acids (FFA) from peripheral fat stores due to enhanced lipolysis, increased de novo hepatocyte triglyceride synthesis from glucose and reduced apo B production, which diminishes fat export from the liver.

In the absence of established treatment, therapy is generally directed to treatment of risk factors for metabolic syndrome. Recently, some studies have been demonstrated that Polyunsaturated fatty acids (PUFAs), omega3 type, could reduced TNFalfa, IL6, aminotransferases, insulin resistance and steatosis verified by ultrasound. Nevertheless, this is the first study that evaluate liver histology after six months of PUFA (omega3) in the treatment of patients with NASH.

Based on these aspects, the aim of this prospective investigation, is evaluate the effectiveness of PUFA (omega3) in the treatment of patients with NASH.

METHODS Population This study will be developed in the center of study of DHGNA/NASH in the Central Institute of the Hospital of the Clinics in São Paulo, Brazil. This study comprised 60 patients diagnosed with NASH based on liver biopsy findings. In addition, all of the patients will have elevated alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) levels on at least two occasions over 6 months prior to enrollment. Other causes of liver disease included a hepatobiliary system ultrasound, viral serology, autoantibody titers, serum iron, ferritin and transferrin saturation, ceruloplasmin and copper levels and alpha1-antitrypsin will be exclude. Patients who have a > 100 g/week alcohol intake determined by a detailed personal history, questioning of family members, and investigation of previous medical records, will be excluded. Patients with steatohepatitis accompanying other liver diseases, or systemic diseases other than obesity, hyperlipidemia, and diabetes or with intake of hepatotoxic drugs or lipid-lowering agents were excluded. Specific informed consent was obtained for the study and the protocol was approved by the Internal Review Board of University of São Paulo. Diagnosis of diabetes type II, hypertension, dyslipidemia were based on the criteria of the American Diabetes Association (fasting glucose above 100mg/dl; Triglyceride > 150mg/dl; HDL < 40mg/dl in man or < 50mg/dl in woman; > 130mmHg systolic or > 85mmHg diastolic)28. Overweight corresponded to body mass index (BMI) ≥ 25 kg/m2 and obesity to BMI ≥ 30 kg/m2.

Study Design Randomized, double blind, placebo controlled. Patients will be randomized into two groups: Group I / control: 30 NASH patients will be receive placebo orally for 6 months Group II /(PUFA-(omega3) : 30 NASH patients will be receive PUFA-(omega3) orally for 6 months

Laboratorial Assays ( every 2 months)

* AST, ALT, FA, GGT, BT/D/I, albumine, INR, plaquettes, Fe, fasting glucose insulin, , peptide C, leptin, Total cholesterol, HDL. LDL, Triglycerides,
* TNFalfa, IL6, adiponectin, lipidic leuckocyte profile, EPA (eicosapentaenoic acid), DHA (docosahexaenoic)

Histological diagnosis Liver tissue will be fixed in 4% formaldehyde and processed for hematoxylin-eosin (HE) and Masson Trichrome stains for histological analysis. All specimens will be scored by a single liver pathologist with expertise in NAFLD: macro- and microvascular fatty change, zonal distribution, foci of necrosis, portal and perivenular fibrosis, and inflammatory and fibrotic infiltrate with zonal distribution. The specimens will be blindly scored according to the NASH Activity Score (NAS) devised by the Pathology Committee of the NASH Clinical Research Network 29. According to the NAS, scored parameters included macro- and microvascular fatty change, zonal distribution, foci of necrosis, portal and perivenular fibrosis, and inflammatory and fibrotic infiltrate with zonal distribution.

ELIGIBILITY:
Inclusion Criteria:

* 18-70 years of age, both sexes
* With or without non-insulin-dependent diabetes or glucose intolerance
* Absence of alcoholism <20g (women) and <40g (men) of ethanol/day, drugs, schistosomiasis, hepatitis B or C and other chronic liver diseases cause determined
* Absence of autoantibodies and rates of copper and ceruloplasmin normal
* Biopsy-liver until 12 months previous, showing steatosis, lobular inflammatory infiltrate and ballooning of hepatocytes, which may be present or not Mallory's corpuscles and liver fibrosis stage I and II, NAS score> 5;
* Patients who agree to participate in the study and all signed informed consent.

Exclusion Criteria:

* Poisoning by exogenous oxidants
* Pregnancy and lactation
* Prothrombin time <70% or platelet count <70 000/mm3, or any bleeding disorders, including alteration of the bleeding time
* Refusal to cooperate with research
* steatosis without signs of inflammation or ballooning or cirrhosis (stage IV)
* diabetes mellitus using insulin
* allergy to fish or flaxseed
* anti-inflammatory use of non-hormonal

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-09; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Efficacy in reduce inflammatory component of NASH for NAS score | 6 months
  Determine the efficacy of Omega-3 fatty acid in reducing the inflammatory component of NASH for liver through liver biopsy NAS score.

SECONDARY OUTCOMES:
Inflammatory systemic profile | 6 mothns
  Measure TNFalfa, IL6, adiponectin, lipidic leuckocyte profile, EPA (eicosapentaenoic acid), DHA (docosahexaenoic) and laboratory tests AST, ALT, Cholesterol, total triglycerides, PCR, VHS, SAA.

CONTACTS AND LOCATIONS:
Overall Officials: CLAUDIA PM OLIVEIRA, MD, PhD, Principal Investigator — University of Sao Paulo, School of Medicine
Locations (1):
- University of Sao Paulo School of Medicine, São Paulo, São Paulo, Brazil